CLINICAL TRIAL: NCT07138768
Title: The Role of MRI in the Early Diagnosis and Management of Acute Stroke and Its Impact on Turnaround Time (TAT) in Emergency Settings
Brief Title: Role of MRI in the Early Diagnosis and Management of Acute Stroke and Its Impact on Turnaround Time in Emergency Settings
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hend Mohammed Mansour, Lecturer of Emergency Medicine and Trauma, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264PR1258/6/25
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Magnetic Resonance Imaging; Diagnosis; Management; Acute Stroke; Turnaround Time; Emergency Settings
MeSH Terms: conditions — Disease; Stroke | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with acute stroke who are admitted to the emergency department.
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Magnetic Resonance Imaging will be performed to all patients

SUMMARY:
This study aims to evaluate the role of stroke protocol in the early diagnosis and management of acute stroke and its effect on turnaround time (TAT) in emergency settings.

DETAILED DESCRIPTION:
Acute stroke is a common and often devastating disorder; however, acute treatments that reduce long-term disability are available if patients present within the time window for treatment.

Computed tomography (CT) or magnetic resonance imaging (MRI) has been used in comprehensive stroke centers, although the role of advanced imaging in the improvement of stroke outcome remains controversial.

MRI offers advantages for the assessment of acute stroke. Changes of acute ischaemic injury are detectable sooner with MRI than with CT, especially with diffusion-weighted imaging, and ischaemic stroke diagnosis with MRI has greater interobserver and intraobserver reliability than CT, even in readers with little experience.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Both sexes.
* Patients with acute stroke who are admitted to the emergency department.

Exclusion Criteria:

* Contraindications to magnetic resonance imaging (MRI) or computed tomography (CT).
* Symptoms strongly suggestive of subarachnoid hemorrhage.
* Initiation of antithrombotic or thrombolytic treatment before the completion of both scans.
* Inability to complete both scans in time to allow thrombolytic treatment within three h of the onset of symptoms.
* Uncontrollable hypertension.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective cohort study will be carried out on 136 patients presenting with acute stroke symptoms after approval from the institutional ethical committee.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2025-08-23 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of magnetic resonance imaging for acute stroke | Immediately post-procedure (Up to 1 hour)
  Sensitivity of magnetic resonance imaging for acute stroke will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.